CLINICAL TRIAL: NCT03946982
Title: Comparisons Between Low Thoracic and Lumbar Epidural Analgesia on Postoperative Pain Management Qualities After Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Comparisons Between Low Thoracic and Lumbar Epidural Analgesia on Postoperative Pain Low Thoracic v.s. Lumbar Epidural for Post-cesarean Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201902009RINC
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2020-05

CONDITIONS: Post-cesarean Pain Control Quality
Keywords: Patient controlled epidural analgesia ,Cesarean delivery,pain management,epidural opioid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low thoracic patient controlled epidural analgesia (Experimental)
  Interventions: Procedure: low thoracic epidural
- Lumbar epidural patient controlled epidural analgesia (Active Comparator)
  Interventions: Procedure: lumbar epidural
- Low thoracic epidural morphine (Active Comparator)
  Interventions: Procedure: low thoracic epidural
- Lumbar epidural morphine (Active Comparator)
  Interventions: Procedure: lumbar epidural

INTERVENTIONS:
Procedure: low thoracic epidural — obstetric epidural catheters inserted at low thoracic intervertebral spaces
  Arms: Low thoracic epidural morphine; Low thoracic patient controlled epidural analgesia
Procedure: lumbar epidural — obstetric epidural catheters inserted at low thoracic intervertebral spaces (conventional)
  Arms: Lumbar epidural morphine; Lumbar epidural patient controlled epidural analgesia

SUMMARY:
Whether low thoracic epidural analgesia improves postoperative cesarean pain qualities than conventional lumbar epidural analgesia?

DETAILED DESCRIPTION:
Postoperative pain remains the leading cause of concern in women faced with undergoing a cesarean delivery. Inadequate acute pain management is associated with numerous negative effects, including delayed postpartum recovery, interference with mother-child bonding because postoperative pain limits breastfeeding, and a high risk of postpartum depression and persistent pain.

Epidural analgesia (EA) is being increasingly preferred to systemic opioid because of better analgesic effect. Although EA is widely used for cesarean delivery, the effect of the site of epidural catheter insertion on the quality of postoperative pain management remains inadequately investigated. For example, placement of the epidural catheter in the low thoracic intervertebral spaces may be more suitable for catheter-incision-congruent analgesia during caesarean delivery than in the lumbar intervertebral space; however, epidural catheter insertion is conventionally recommended at the lumbar intervertebral space. Therefore, in this study, we aim to investigate the difference in post-cesarean pain control quality between low thoracic EA and lumbar EA.

ELIGIBILITY:
Inclusion:

1. age between 20-yr and 50-yr parturients
2. elective cesarean delivery

Exclusion:

1. contraindicated to regional anesthesia, eg. coagulopathy (INR> 1.5; platelet< 80000...etc)
2. significant co-morbidities, eg. preeclamspia, heart failure with New York Heart Association (NYHA) Classification> class 2
3. allergy to opioids or local anesthetics

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women with a visual analogue scale> 33 mm | postoperative two days
Pain intensity | postoperative two days
  pain intensities in three category, namely static, dynamic and uterine cramping, gauged by a 100 mm visual analogue scale

SECONDARY OUTCOMES:
Adverse effects | postoperative two days
  Incidences of epidural-related adverse effects including sedation states, sensory blockade, motor blockade, pruritus, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan